CLINICAL TRIAL: NCT01214681
Title: Chemoprevention of Colorectal Cancer: the Role of Non-digestible Carbohydrates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Newcastle University (Other)
Collaborators: Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 002
Record Dates: First submitted 2010-10-01; First posted 2010-10-05 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Colorectal Cancer
Keywords: Biomarkers; Colorectal cancer; Resistant starch; Polydextrose; Non-digestible carbohydrate
MeSH Terms: conditions — Colorectal Neoplasms | interventions — maltodextrin; high-amylose maize type 2 resistant starch, maize; polydextrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin and Amioca starch
- Hi-maize 260 (Experimental)
  Interventions: Dietary Supplement: Hi-maize 260
- Polydextrose (Experimental)
  Interventions: Dietary Supplement: Polydextrose
- Hi-maize 260 and polydextrose (Active Comparator)
  Interventions: Dietary Supplement: Hi-maize 260 and polydextrose

INTERVENTIONS:
Dietary Supplement: Maltodextrin and Amioca starch — 12g Maltodextrin and 23g Amioca starch daily in divided doses for 50 days. Provided as a powder to be added to food or drink.
  Arms: Placebo
Dietary Supplement: Hi-maize 260 — 23g Hi-maize 260 and 12g Maltodextrin daily in divided doses for 50 days. Provided as a powder to be added to food or drink.
  Arms: Hi-maize 260
Dietary Supplement: Polydextrose — 12g polydextrose and 23g amioca starch daily in divided doses for 50 days. Provided as a powder to be added to food or drink.
  Arms: Polydextrose
Dietary Supplement: Hi-maize 260 and polydextrose — 12g polydextrose and 23g Hi-maize 260 daily in divided doses for 50 days. Provided as a powder to be added to food or drink.
  Arms: Hi-maize 260 and polydextrose

SUMMARY:
Colorectal cancer is a common disease worldwide. It is now thought that colorectal cancer cells arise from stem cells where the genetic material regulating growth and division of the stem cell has become defective. This leads to unregulated production of cells which in turn have defective genetic information and cancer formation.

Research into colorectal cancer is hampered by the fact that studies must take a very long time to produce results and be very large if the development of a cancer is the endpoint. Therefore alternative methods of quantifying the risk of developing a cancer are required so trials can be a realistic size and be completed in a realistic time frame. The investigators have previously identified several candidates for these 'biomarkers'. The next stage in proving or disproving these as useful biomarkers is to test their response to a dietary agent that the investigators know reduces the risk of colon cancer.

DETAILED DESCRIPTION:
This project is designed to enhance understanding of links between food and the health of the gut. The particular purpose of the project is to investigate the impact of a well-defined intervention in human volunteers on a panel of novel, and established, diet-related biomarkers of bowel cancer risk. We have developed a number of novel biomarkers of diet-related CRC risk measured in colo-rectal mucosal biopsies (and in stool). These biomarkers include differentially expressed proteins, DNA methylation markers and inflammation markers. In our on-going BORICC Study we are investigating the relationships between dietary exposure and nutritional status for these biomarkers in a cross-sectional study. The next logical step in this research is to determine whether a selected panel of the most promising biomarkers responds to a dietary intervention i.e. to test their utility as biomarkers of GI health and potential as surrogate endpoints in future human studies.

We propose to use Hi-maize 260 and polydextrose (PD) as our model resistant starch (RS) intervention agents. RS describes the fraction of dietary starch which is not digested in the small bowel and which flows to the colon where it is a substrate for bacterial fermentation. (Asp, 1996) PD is produced by the bulk melt polycondensation of glucose and sorbitol to produce an oligosaccharide with a mean degree of polymerisation of 12 which is resistant to mammalian GI enzymes and, like other RSs, is a substrate for bacterial fermentation. (Auerbach, 2007) Both Hi-maize and PD are fermented (to a greater or lesser extent) producing short-chain fatty acids (SCFA) including butyrate. (Asp, 1996) Butyrate has beneficial effects on gut physiology and immune function including anti-inflammatory effects. (Wächtershäuser, 2000; Dronamraju, 2009)

In the present project we will investigate the impact of PD and RS, as food-borne substrates for delivery of butyrate, on biomarkers of bowel cancer risk.

ELIGIBILITY:
Inclusion Criteria:

Attended for flexible sigmoidoscopy or colonoscopy and no macroscopic pathology identified

Exclusion Criteria:

* Age <16 or >85
* Familial polyposis syndrome
* Lynch syndrome
* Known colorectal tumour
* Previous colorectal resection
* Pregnancy
* Chemotherapy in last 6 months
* Therapy with aspirin/other NSAID
* Other immunosuppressive medication
* Active colonic inflammation at endoscopy
* Incomplete left sided examination
* Colorectal carcinoma found at endoscopy
* Iatrogenic perforation at endoscopy
* Colorectal cancer on histology
* Warfarin or other anticoagulant use
* Diabetes mellitus
* Crohn's disease
* Cognitive impairment

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Faecal calprotectin concentration | 50 days

SECONDARY OUTCOMES:
Serum C reactive protein concentration | 50 days
COX 2 expression in mucosal biopsies | 50 days
Number and distribution of mitotic and apoptotic cells within colonic crypts (mucosal cell kinetics) | 50 days
Cellular CDK 4 RNA expression | 50 days
Cellular GADD45A RNA expression | 50 days
Target gene methylation (p16, GSTP1, RARβ2, CDH1 GATA4 APC, SFRP1, 2, 4 and 5, AXIN2, DKK1 and WIF1) | 50 days
Global genetic methylation | 50 days
Cellular protein biomarker (CK8) expression | 50 days
Faecal pH | 50 days
Faecal bacterial abundance and population | 50 days
Faecal short chain fatty acid concentration | 50 days
Urinary short chain fatty acid concentration | 50 days
Plasma short chain fatty acid concentration | 50 days

CONTACTS AND LOCATIONS:
Overall Officials: John Mathers, PhD, Study Director — Newcastle University; Naomi Willis, PhD, Principal Investigator — Newcastle University
Locations (2):
- United Kingdom (2):
  - Wansbeck General Hospital, Ashington, Northumberland
  - North Tyneside General Hospital, North Shields, Tyne & Wear

REFERENCES:
- [Result] Asp NG, van Amelsvoort JM, Hautvast JG. Nutritional implications of resistant starch. Nutr Res Rev. 1996 Jan;9(1):1-31. doi: 10.1079/NRR19960004. No abstract available. PMID 19094263
- [Result] Auerbach MH, Craig SA, Howlett JF, Hayes KC. Caloric availability of polydextrose. Nutr Rev. 2007 Dec;65(12 Pt 1):544-9. doi: 10.1301/nr.2007.dec.544-549. PMID 18236693
- [Result] Wachtershauser A, Stein J. Rationale for the luminal provision of butyrate in intestinal diseases. Eur J Nutr. 2000 Aug;39(4):164-71. doi: 10.1007/s003940070020. PMID 11079736
- [Result] Dronamraju SS, Coxhead JM, Kelly SB, Burn J, Mathers JC. Cell kinetics and gene expression changes in colorectal cancer patients given resistant starch: a randomised controlled trial. Gut. 2009 Mar;58(3):413-20. doi: 10.1136/gut.2008.162933. Epub 2008 Oct 31. PMID 18978177
- [Derived] Malcomson FC, Willis ND, McCallum I, Xie L, Lagerwaard B, Kelly S, Bradburn DM, Belshaw NJ, Johnson IT, Mathers JC. Non-digestible carbohydrates supplementation increases miR-32 expression in the healthy human colorectal epithelium: A randomized controlled trial. Mol Carcinog. 2017 Sep;56(9):2104-2111. doi: 10.1002/mc.22666. Epub 2017 May 9. PMID 28418082
- [Derived] Malcomson FC, Willis ND, McCallum I, Xie L, Ibero-Baraibar I, Leung WC, Kelly S, Bradburn DM, Belshaw NJ, Johnson IT, Mathers JC. Effects of supplementation with nondigestible carbohydrates on fecal calprotectin and on epigenetic regulation of SFRP1 expression in the large-bowel mucosa of healthy individuals. Am J Clin Nutr. 2017 Feb;105(2):400-410. doi: 10.3945/ajcn.116.135657. Epub 2017 Jan 11. PMID 28077379